CLINICAL TRIAL: NCT02057744
Title: Multi-center, Partially Randomized, Controlled Trial of MIS Robotic vs. Freehand in Short Adult Degenerative Spinal Fusion Surgeries
Brief Title: MIS ReFRESH: Robotic vs. Freehand Minimally Invasive Spinal Surgeries
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mazor Robotics (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN110
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Degenerative Spine Disease; Spondylolisthesis; Spondylosis
Keywords: Robotic-guided surgery; Minimally invasive spinal surgery; Spinal fusion; Pedicle screws
MeSH Terms: conditions — Spondylolisthesis; Spondylosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Robotic-guided: Adult patients (21 years or older) undergoing short (4 or less consecutive vertebrae) thoracic, lumbar or lumbosacral percutaneous/minimally invasive robotic-guided spinal fixation surgery.
- Freehand image-guided: Adult patients (21 years or older) undergoing short (4 or less consecutive vertebrae) thoracic, lumbar or lumbosacral percutaneous/minimally invasive image-guided freehand or navigated spinal fixation surgery.

SUMMARY:
To quantify potential short- and long-term benefits of robotically-guided minimally invasive spine surgery (MIS) for adult patients with lower back degeneration, in comparison a matching group of control patients operated in a minimally invasive approach whether freehand or with image guidance or navigation techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age over 21 years), undergoing short (4 or less consecutive vertebrae) lumbar or lumbosacral percutaneous/MIS spinal fixation surgery.
2. May include surgeries involving iliac screws, although these screws will not be included in the data analysis.
3. Primary fusion surgery
4. Patient capable of complying with study requirements
5. Signed informed consent by patient

Exclusion Criteria:

1. Pregnancy
2. Revision surgery (prior laminectomy or discectomy is not excluded).
3. Infection or malignancy
4. Primary abnormalities of bones (e.g. osteogenesis imperfecta)
5. Primary muscle diseases, such as muscular dystrophy
6. Neurologic diseases (e.g. Charcot-Marie Tooth, Guillain-Barre syndrome, cerebral palsy, spina bifida or neurofibroma)
7. Spinal cord abnormalities with any neurologic symptoms or signs
8. Spinal cord lesions requiring neurosurgical interventions, such as hydromyelia
9. Paraplegia
10. Patients who have participated in a research study involving an investigational product in the 12 weeks prior to surgery
11. Patients requiring anterior release or instrumentation
12. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study.
13. Patient cannot follow study protocol, for any reason
14. Patient cannot or will not sign informed consent

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (21 years or older) undergoing short (4 or less consecutive vertebrae) thoracic, lumbar or lumbosacral percutaneous/minimally invasive spinal fixation sugery.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2014-10; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Intra-operative exposure to x-ray radiation | Day of surgery
  Reading of exposure in seconds (and KvP if available) from C-arm or other imaging system used in the operating room.
Surgical complications | Within first year from day of surgery
  New neural deficits, implant-related durotomy, infection requiring return to surgery, hardware failure requiring removal, vertebral body fracture, failure to fuse
Revision surgeries | 1 year
  All cause revisions

SECONDARY OUTCOMES:
Pedicle screw instrumentation accuracy | Within 1 year of surgery, if indicated by surgeon and clinically necessary
  Accuracy will be quantified in millimeters and scored using the Gertzbein-Robbins classification, based on postoperative CTs that are clinically necessary for the management of the patient.
Incidence of pseudoarthrosis (malunion) | Within 1 year from surgery
  Failure of the operated spinal segment to fuse.
Length of convalescence | Within 1 year of surgery
  Length of stay at the hospital, destination at discharge, time to return to normal activities, time to return to work
Times of intra-operative stages | Day of surgery
  instrumentation time per screw, total surgery time
Ratio of executed vs. planned screws | Day of surgery
  number of screws planned to be robotically inserted and manually inserted instead and cause.
Quality of life assessment | Each visit up to 1 year1
  Health related quality of life questionnaires, including: back and leg Visual Analog Scale (VAS), Oswestry Disability Index (ODI), European Quality % Dimensions (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Doron Dinstein, MD, Study Director — Mazor Robotics, Ltd
Locations (9):
- United States (9):
  - Florida Hospital Celebration Health, Celebration, Florida
  - Baptist Health, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Central Florida Neurosurgery Institute, Orlando, Florida
  - Southeastern Spine Center & Research Institute, Sarasota, Florida
  - The Rothman Institute, Abington, Pennsylvania
  - Tabor Orthopedics, Memphis, Tennessee
  - Atlantic Brain & Spine, Fairfax, Virginia
  - Virginia Spine Institute, Reston, Virginia

REFERENCES:
- [Background] Devito DP, Kaplan L, Dietl R, Pfeiffer M, Horne D, Silberstein B, Hardenbrook M, Kiriyanthan G, Barzilay Y, Bruskin A, Sackerer D, Alexandrovsky V, Stuer C, Burger R, Maeurer J, Donald GD, Schoenmayr R, Friedlander A, Knoller N, Schmieder K, Pechlivanis I, Kim IS, Meyer B, Shoham M. Clinical acceptance and accuracy assessment of spinal implants guided with SpineAssist surgical robot: retrospective study. Spine (Phila Pa 1976). 2010 Nov 15;35(24):2109-15. doi: 10.1097/BRS.0b013e3181d323ab. PMID 21079498
- [Background] Kantelhardt SR, Martinez R, Baerwinkel S, Burger R, Giese A, Rohde V. Perioperative course and accuracy of screw positioning in conventional, open robotic-guided and percutaneous robotic-guided, pedicle screw placement. Eur Spine J. 2011 Jun;20(6):860-8. doi: 10.1007/s00586-011-1729-2. Epub 2011 Mar 8. PMID 21384205
- [Background] Hu X, Ohnmeiss DD, Lieberman IH. Robotic-assisted pedicle screw placement: lessons learned from the first 102 patients. Eur Spine J. 2013 Mar;22(3):661-6. doi: 10.1007/s00586-012-2499-1. Epub 2012 Sep 14. PMID 22975723